CLINICAL TRIAL: NCT05350462
Title: ADOPT - Community Intervention: Social Science Research Study to Support the Adoption of Levo-Praziquantel (L-PZQ) for the Treatment of Schistosomiasis in Pre-school Aged Children in Côte d'Ivoire, Kenya and Uganda
Brief Title: Adoption of L-PZQ for Schistosomiasis by Endemic Counties - Social Science Research Study
Acronym: ADOPT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: African Institute for Health and Development (Unknown); Makerere University (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Global Health Innovative Technology Fund (Other); Stichting Lygature (Unknown); Université Félix Houphouët-Boigny (Unknown); Kenya Medical Research Institute (Other); Swiss Tropical & Public Health Institute (Other); SCI Foundation (Unknown)
Responsible Party: Principal Investigator, Andrea Winkler, Prof. Dr. Dr., Technical University of Munich
Other Study IDs: 731/21 S; RIA2019IR-2895 (Other Grant/Funding Number: EDCTP); G2020-102R1 (Other Grant/Funding Number: GHIT)
Record Dates: First submitted 2022-04-14; First posted 2022-04-28 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Schistosomiasis in Children; Social Acceptance
Keywords: key informant interview; mixed methods; qualitative research; focus group discussion; neglected tropical diseases; community health; pre-school aged children; Sub-Saharan Africa; Kenya; Uganda; Ivory Coast; Public-private partnership; collaborative research; implementation study; social acceptance; levo-praziquantel; mass drug administration; Côte d'Ivoire; knowledge; health literacy
MeSH Terms: conditions — Neglected Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Agboville, Côte d'Ivoire: Drug naive region
  Parents/guardians of pre-school aged children Primary healthcare personnel Community stakeholders (e.g. political/administrative leaders, religious leaders, traditional healers, civil society, non-governmental organizations, key health system representatives, schistosomiasis control officers, community drug distributers)
  Interventions: Behavioral: Community pilot L-PZQ distribution - intervention is NOT part of this observational study
- Bangolo, Côte d'Ivoire: Drug naive region
  Parents/guardians of pre-school aged children Primary healthcare personnel Community stakeholders (e.g. political/administrative leaders, religious leaders, traditional healers, civil society, non-governmental organizations, key health system representatives, schistosomiasis control officers, community drug distributers)
- Man, Côte d'Ivoire: was a phase III clinical trial site for Levo-Praziquantel in 2021
  Parents/guardians of pre-school aged children Primary healthcare personnel Community stakeholders (e.g. political/administrative leaders, religious leaders, traditional healers, civil society, non-governmental organizations, key health system representatives, schistosomiasis control officers, community drug distributers)
  Interventions: Behavioral: Community pilot L-PZQ distribution - intervention is NOT part of this observational study
- Homa Bay, Kenya: was a phase III clinical trial site for Levo-Praziquantel in 2021
  Parents/guardians of pre-school aged children Primary healthcare personnel Community stakeholders (e.g. political/administrative leaders, religious leaders, traditional healers, civil society, non-governmental organizations, key health system representatives, schistosomiasis control officers, community drug distributers)
  Interventions: Behavioral: Community pilot L-PZQ distribution - intervention is NOT part of this observational study
- Kwale, Kenya: Drug naive region
  Parents/guardians of pre-school aged children Primary healthcare personnel Community stakeholders (e.g. political/administrative leaders, religious leaders, traditional healers, civil society, non-governmental organizations, key health system representatives, schistosomiasis control officers, community drug distributers)
  Interventions: Behavioral: Community pilot L-PZQ distribution - intervention is NOT part of this observational study
- Hoima, Uganda: Drug naive region
  Parents/guardians of pre-school aged children Primary healthcare personnel Community stakeholders (e.g. political/administrative leaders, religious leaders, traditional healers, civil society, non-governmental organizations, key health system representatives, schistosomiasis control officers, community drug distributers)
  Interventions: Behavioral: Community pilot L-PZQ distribution - intervention is NOT part of this observational study
- Bugiri, Uganda: Drug naive region
  Parents/guardians of pre-school aged children Primary healthcare personnel Community stakeholders (e.g. political/administrative leaders, religious leaders, traditional healers, civil society, non-governmental organizations, key health system representatives, schistosomiasis control officers, community drug distributers)
  Interventions: Behavioral: Community pilot L-PZQ distribution - intervention is NOT part of this observational study

INTERVENTIONS:
Behavioral: Community pilot L-PZQ distribution - intervention is NOT part of this observational study — Data collection will occur at two main time points of the ADOPT-community intervention project: before (baseline assessment) and during/after the community pilot L-PZQ distribution, in order to inform the design and process of the implementation, including that of advocacy and mobilisation, of Levo-Praziquantel delivery to PSAC.
  Groups: Agboville, Côte d'Ivoire; Bugiri, Uganda; Hoima, Uganda; Homa Bay, Kenya; Kwale, Kenya; Man, Côte d'Ivoire

SUMMARY:
Knowledge, acceptability and perception of paediatric schistosomiasis and its treatment will be explored through a social science-driven mixed-methods approach within three endemic countries: Kenya, Uganda and Côte d'Ivoire.

DETAILED DESCRIPTION:
In many African countries, the worm disease schistosomiasis, also known as bilharzia, is a serious problem that affects the health of many people. An estimated 50 million pre-school children in sub-Saharan Africa are affected, but are currently excluded from routine preventive chemotherapy with praziquantel because there is no suitable preparation for this age group. As a result, the public-private Pediatric Praziquantel Consortium, led by the pharmaceutical company Merck, has developed Levo-Praziquantel 150 mg, which is child-friendly in dosage as well as in tolerability and taste. The European & Developing Countries Clinical Trials Partnership (EDCTP) programme, together with the Global Health Innovation Technology Fund (GHIT), is funding the conduct of an implementation study "ADOPT - Adoption of Levo-Praziquantel 150mg for Schistosomiasis by endemic countries" to prepare for the introduction of Levo-Praziquantel in the partner countries Kenya, Côte d'Ivoire and Uganda, where schistosomiasis is endemic.

This study protocol describes the social science research part of the implementation project (Work Package 1). It aims to provide important insights into local conditions as well as knowledge, perceptions and management of schistosomiasis among the population in each of the three study countries, particularly among parents of young children and health workers. In addition, possible factors influencing the introduction and acceptance of the new preparation will be identified, as well as ideal platforms for this. Furthermore, the implementation pilot study will be accompanied and its implementation investigated.

The mixed-methods study with a focus on qualitative research methods will be conducted in two different phases in the three partner countries: 1) before the intervention/pilot study; 2) during and after the implementation pilot study. In the first phase, semi-structured Key Informant Interviews (KIIs) will be conducted with health workers and stakeholders from the Neglected Tropical Diseases (NTD) sector and local health workers in the study regions. In addition, parents/families of young children will be interviewed through focus group interviews (FGD) and socio-demographic questionnaires. Study design, data collection and analysis as well as publication and dissemination are carried out jointly by the social science research team of the TUM Center for Global Health and the partners in the study countries.

The formative qualitative evaluation of the post-intervention part will be conducted after the community pilot Levo-Praziquantel distribution (which is not part of this observational study) with the same key informants as preADOPT intervention. This will entail documentation of implementation strategies on the ground through participant observations, semi-structured and in-depth interviews and FGDs to assess the realisation and acceptance of the different strategies. We will also add a new key informant group, i.e. community drug distributors, of which participants will be recruited into semi-structured and in-depth interviews as well as FGDs. For the post-intervention, the same methods as described above for preintervention will be applied. In addition, a postintervention simple questionnaire will be added to the parent/guardian group (designed on the basis of findings from the pre-intervention part) to assess the implementation process.

ELIGIBILITY:
Inclusion Criteria:

* within the targeted communities
* all key informant groups as described
* willing to participate voluntarily and to provide informed consent

Exclusion Criteria:

- refusing to give informed consent, participating not voluntarily or their participation causing psycho-social distress or even harm to themselves or other community members

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study populations will consist of key informants, such as parents/guardians of PSAC, frontline health personnel, community and religious leaders, key healthcare workers, community health stakeholders and schistosomiasis control officials, in each study site in each of the three countries. Selection and recruitment of participants for qualitative interviews will be purposive.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative data analysis including self-reported information on knowledge, perception, and experience of schistosomiasis (treatment) and child health within families (Micro, Meso and Macro level) | 13.12.2021 -31.06.2022 + Second study wave in 2024
  Qualitative data analysis using the "Thematic Analysis" approach. This approach helps to identify, analyse and interpret patterns of meaning in the form of emerging "themes" in the qualitative data. Important "themes" emerging from the focus group discussions and key informant interviews are explored.
  In this way, important subjective factors of acceptance or non-acceptance as well as differences within opinions can be revealed. Topics on which the qualitative analysis will focus are:
  * Characterization and summary of knowledge, experience and views of parents/guardians of PSAC as well as health care providers and health authorities about schistosomiasis and its treatment. Comparison across study sites and countries.
  * Comparison of data, which is collected prior to the intervention, and data collected during/after the intervention.
Semi-structured socio-demographic questionnaires (quantitative data) used to collect further data from parents/guardians of PSAC in the study (knowledge, perception and acceptability related to (pediatric) schistosomiasis) | 13.12.2021 -31.06.2022 + Second study wave in 2024
  The outcomes of the quantitative da will be triangulated with qualitative data (Outcome 1) and secondary data from a desk review.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Nyamongo, Dr., Principal Investigator — African Institute for Health and Development; Stella Neema, Prof., Principal Investigator — Makerere University - Social Science Department; Alain Toh, Prof., Principal Investigator — Université Félix Houphouët-Boigny d'Abidjan-Cocody
Locations (3):
- Université Félix Houphouët-Boigny, Abidjan, Côte d’Ivoire
- African Institute for Health and Development, Nairobi, Kenya
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers in order to protect their privacy. Anonymised data will be available upon request.